CLINICAL TRIAL: NCT03050580
Title: An Evaluation of the "Treatment Group Model for Abused Women" in Shelters in Hong Kong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Anna W.M. Choi, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW12-557
Record Dates: First submitted 2017-02-01; First posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Abused Women
Keywords: Abused women; treatment group; family violence
MeSH Terms: interventions — Standard of Care; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-esteem enhancement group (Experimental): The self-esteem enhancement group service for abused women will receive a six-session program for recognizing strengths and resources through group activities and sharing.
  Interventions: Behavioral: self-esteem enhancement group
- Standard care (Active Comparator): The shelter standard care for abused women includes residential accommodations, emotional support, legal, housing and financial advice and referral service.
  Interventions: Behavioral: Standard care for abused women

INTERVENTIONS:
Behavioral: self-esteem enhancement group — Subjects in the treatment group will join a six-session treatment for recognizing their strengths and resources through group activities and sharing. Each session is 1.5-2 hours long, and all sessions are designed for 4-8 abused women. The activities are designed and led with an aim to improve their self-esteem, general health, as well as to reduce the level of depression. This service is provided by registered social workers.
  Other Names: experimental/treatment group
  Arms: Self-esteem enhancement group
Behavioral: Standard care for abused women — The shelter standard care and services will be provided to the abused women in one randomized shelter. Besides, standard care in shelters includes residential accommodations, emotional support, legal, housing and financial advice and referrals will be given to survivors who reported being abused.
  Other Names: control group
  Arms: Standard care

SUMMARY:
This is cluster randomized control trial, that aims to evaluate the effectiveness of the treatment group model for abused women in enhancing their self-esteem and reducing the level of depression, in three shelters for abused women of Po Leung Kuk (a social service organization in Hong Kong). It is hypothesized that subjects in the Treatment Group would report significant improvement in self-esteem, social support, quality of life; reduction in the level of depression, symptoms of Posttraumatic Stress Disorder at 3 months after service delivery.

DETAILED DESCRIPTION:
This is cluster randomized control trial, that aims to evaluate the effectiveness of the treatment group model for abused women in enhancing their self-esteem and reducing the level of depression, in three shelters for abused women of Po Leung Kuk (a social service organization in Hong Kong). 50-60 abused women are recruited as treatment group from two randomized shelters of Po Leung Kuk (Shelters A and B), where subjects receive self-esteem enhancement group intervention for abused women. Another 50-60 abused women are recruited as the control group from a randomized shelter of Po Leung Kuk (Shelter C), where subject receive standard shelter services for abused women. It is hypothesized that subjects in the Treatment Group would report significant improvement in self-esteem, social support, quality of life; reduction in the level of depression, symptoms of Posttraumatic Stress Disorder at 3 months after service delivery, are compared to those in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Abused women of family violence aged 18 or older
* Receiving services from shelters of Po Leung Kuk

Exclusion Criteria:

* Unable to communicate (possible reasons: dialects used by targets but not understandable by interviewers; mentally challenged)
* Unable to give consent to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Changes of self-esteem from baseline to 3 months | Baseline; 3 months
  Confidence in one's own worth or abilities; self-respect; feeling of powerlessness.
  Rosenberg Self-Esteem Scale (Rosenberg, 1965) will be used to measure the self-esteem of the participants. This is a 10-item Likert-type scale on a 4-point scale ranging from strongly agree to strongly disagree. The scores for the 10 items are then summed; the higher the score, the higher the participant's self-esteem.

SECONDARY OUTCOMES:
Basic demographics data questionnaire | Baseline
  Basic demographics data: Age, ethnicity, marital status, living arrangements with spouse/partner, education level, occupation, immigration status (if applicable), information on support network (family and friend), action plan (e.g., filing divorce, application of Injunctions)
Social support | Baseline; 3 months
  Self-perceived social support from others
  The Interpersonal Support Evaluation List-12 (ISEL-12) (Cohen et al., 1985), will be used to measure social support. It has has good psychometric properties and good internal consistency (Cronbach α = 0.88), was used to measure the perceived social support of abused women. The 12-item questionnaire measures 3 sub-scales consisting of appraisal, belonging and tangible support, each of which has 4 items. Each item scores from 0 (definitely false) to 3 (definitely true) giving a total score ranging from 0 to 36. The higher the score, the more the women perceive that they received social support.
Level of depression | Baseline; 3 months
  Self-report symptoms corresponding to criteria for diagnosing depressive disorders
  The Beck Depression Inventory version II (BDI-II) will be used to measure level of depression. It is a self-report instrument for the assessment of symptoms corresponding to criteria for diagnosing depressive disorders (Beck, Steer, & Brown, 1996). It consists of 21 groups of statements and requires the respondent to choose one statement in each group that best describes her during the previous two weeks. The BDI-II has been translated into Chinese and has demonstrated satisfactory validity and reliability (α ranged from .86 to .87) (Leung, 2001).
Post-traumatic Stress Disorder symptoms | Baseline; 3 months
  Self-report symptoms corresponding to criteria for diagnosing Post-traumatic Stress Disorder symptoms
  The Chinese Version of the Impact of Event Scale-Revised (IES-R) (Chen et al., 2005 Wu and Chan, 2003) will be used to assess the PTSD symptoms of participants. This is a 22-items self-report instrument to assess PTSD symptoms after a specific traumatic stressor. There are three subscales, including intrusive, avoidance, and hyperarousal symptoms, corresponding to the three dimensions of the DSM-IV criteria for PTSD (American Psychiatric Association, 1994). Each participant will be asked to indicate the frequency of their distress for each of the 22 items on four point scale (0=not at all, 1=seldom, 3=sometime, 4=often).
Quality of life | Baseline; 3 months
  Health-related quality of life
  The SF-12 - Short Form Health Survey (SF-12) will be used to assess health-related quality of life (Ware, Snow & Kosinski, 1993). It consists of 36 items with one measuring health transition and the remaining 35 grouped under eight scales: physical functioning (PF), role limitation due to physical health problems (role-physical; RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role limitation due to emotional health problems (role-emotional; RE) and mental health (MH).
Spousal violence | Baseline; 3 months
  Spousal violence includes any form of physical, psychological and sexual abuse between experienced by the abused women.
  The Chinese version of the Abuse Assessment Screen (C-AAS) will be used to assess participants for IPV. The C-AAS addresses physical, psychological and sexual abuse. The main difference between the original AAS for women (McFarlane, Parker, Soeken & Bullock, 1992) and the C-AAS is that the C-AAS addresses emotional and physical abuse separately in both lifetime and the preceding 3 months while the English AAS measures psychological and physical abuse simultaneously for the lifetime period.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Choi, PhD, Principal Investigator — annachoi@socwork.hku.hk

IPD SHARING:
Plan to Share IPD: Undecided